CLINICAL TRIAL: NCT06748482
Title: Effect of Clinical Pharmacist Consultation on Pain Management Following Pacemaker Implantation
Brief Title: Effect of Clinical Pharmacist Consultation on Pain Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anwar Mohsen Naji Bin Ali Alhaj (Other)
Responsible Party: Sponsor-Investigator, Anwar Mohsen Naji Bin Ali Alhaj, Principal investigator, clinical pharmacist, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pain management by pharmacists
Record Dates: First submitted 2024-12-14; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Pacemaker; Pain Management
Keywords: clinical pharmacist; pain management; pacemaker implantation
MeSH Terms: conditions — Agnosia | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): Will receive standard care for post pacemaker implantation surgery which include a physician interview giving the advice and restrictions regarding the proper position of the left hand and the activities that should be avoided, in addition, a printed paper includes the medication with their doses and the advice that was given orally by the physician
- Intervention group (Other): patients will receive standard care for post PM implantation surgery plus clinical pharmacist consultation through direct interview on day 0 pre-discharge and by telephone on days 1 and 7 post discharge a 15-minute-consultation session with the clinical pharmacist will include detailed and personalized advice on how each patient should take his prescribed medications, the best time to take them, the possible drug-drug interactions, the possible adverse effects such as post operative nausea and vomiting (PONV), bleeding, fever and infection and the required action. A written paper outlining the main points including the detailed protocol with times and doses will be handed to the patient at the end of the consultation. Moreover, a recorded voice note with the detailed protocol will be sent to the patients via the WhatsApp application
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Behavioral: Counseling — a 15-minute-consultation session with the clinical pharmacist will include detailed and personalized advice on how each patient should take his prescribed medications, the best time to take them, the possible drug-drug interactions, the possible adverse effects such as post operative nausea and vomiting (PONV), bleeding, fever and infection and the required action. A written paper outlining the main points including the detailed protocol with times and doses will be handed to the patient at the end of the consultation. Moreover, a recorded voice note with the detailed protocol will be sent to the patients via the WhatsApp application
  Arms: Intervention group

SUMMARY:
This study aims to evaluate the effects of clinical pharmacists' consultation on patients' pain management following Pacemaker implantation surgery.

DETAILED DESCRIPTION:
During the study period, a total of 60 patients who had PM implantation surgeries will be recruited.

• Patients who had PM implantation surgeries in the Mabarra Heart Academy (MHA) will be randomly distributed into two groups using the sealed envelope randomization program: Control group : (30) patients will receive standard care for post pacemaker implantation surgery Intervention group : (30) patients will receive standard care for post PM implantation surgery plus clinical pharmacist consultation through direct interview on day 0 pre-discharge and by telephone on days 1 and 7 post discharge.

* On day 0 pre-discharge, patients' characteristics and medical history will be collected. In addition, patients' quality of life (QoL) will be assessed using European QoL 5-Dimentions 5-Levels version (EQ-5D-5L) - a Patient Reported Outcome (PRO) test that asks five questions to assess patients' overall quality of life, regardless of their medical problems- which contains a vertical EQ visual analog scale (EQ VAS, 0-100 points) and a descriptive EQ-5D-5L system. where the best possible health status is represented by an index value of 1, while the worst possible health state is represented by an index value of <0 . The instructions on how to fill the questionnaire will be explained to the patients and the questionnaire will be self-administered before the operation and two copies of the questionnaire will be given to them to be self-administered at home. Furthermore, pain scores will be assessed using numeric pain rating scale; patients will rate their pain on a scale from 0 to 10, where 0 indicates no pain and 10 indicates intolerable pain. All patients will be given a printed visual pain score to use to report their pain score daily.
* For both groups, pain scores will be reported daily via a WhatsApp message. In addition, on days 1 and 7, patients' QoL will be assessed as the researcher will remind the patients during the phone calls to fill the self-administered questionnaires at home on days 1 and 7. The photos of the answered questionnaires will be afterwards sent to the researcher via the WhatsApp application and the hardcopies will be collected from the patients later on day 10. Furthermore, the presence of any other side effects and the number of times they have contacted their physicians will be reported.
* For the intervention group on day 0; a 15-minute-consultation session with the clinical pharmacist will include detailed and personalized advice on how each patient should take his prescribed medications, the best time to take them, the possible drug-drug interactions, the possible adverse effects such as post operative nausea and vomiting (PONV), bleeding, fever and infection and the required action. A written paper outlining the main points including the detailed protocol with times and doses will be handed to the patient at the end of the consultation. Moreover, a recorded voice note with the detailed protocol will be sent to the patients via the WhatsApp application. They will be told that the researcher will contact them by telephone on days 1 and 7 to follow up with them and collect some information.
* For the control group on day 0; they will be told to contact their physician in case they have any questions or suffer from any adverse effects. They will be told that the researcher will contact them by telephone on days 1 and 7 to collect some information only.
* For the intervention group on day 1 and day 7 post-operation, direct communication by telephone will be conducted. Patients' adherence to their prescriptions will be assessed on a five-point scale where 5 = never, 4 = rarely, 3 = sometimes, 2 = often and 1 = always. Scores will be summed to give a total score, with higher scores indicating higher levels of reported adherence and they will be encouraged to adhere to their medications. Adverse effects will be recorded and recommendation on how to manage them -if present- will be explained. In addition, complications or signs of wound infection such as fever or redness or any other events related to the surgery will be reported and, in such case, patients will be advised to contact their physician.
* On day 10 post operation, a direct interview will be conducted for both groups to assess patients' outcomes in terms of pain severity, medication adherence by tablet counting method, the percentage of patients with unresolved side effects and wound infections, patients' QoL by the self-administered questionnaire, how many times they contacted their physician and the level of patients' satisfaction with medical services. Patient's satisfaction will be assessed using the short assessment of patients' satisfaction (SAPS) which is a seven questions survey with a score range of 0 to 28 where 0 indicates extremely dissatisfied and 28 indicates extremely satisfied

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone pacemaker implantation surgery.
* Patients > 18 years.
* The availability of smartphone with the patient or his caregiver with WhatsApp service on it.

Exclusion Criteria:

* Patients with a history of chronic pain.
* Patients on long-term analgesic therapy.
* Patients suffering from cognitive impairment or psychiatric disorders.
* Pregnant women.
* Patients experiencing surgical complications that may interfere with pain assessment.
* Patients who refuse to participate in the study.
* Illiterate patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-04 (Estimated); Primary Completion 2025-06-24 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Painful episodes, Medication adherence, Wound infection, Quality of life, Adverse effects | 11 days from day 0 (the day of the operation) to day 10 post operation
  Painful episodes: the percentage of patients exhibiting one or more painful episodes of a pain score more than three on a numeric scale from 0 to 10, at days from 1 to 10 throughout the follow-up period.
  Medication adherence: the percentage of patients' adherent to their prescriptions as recommended.
  Wound infection: the percentage of patients who experienced a wound infection at the site of PM insertion.
  QoL: the percentage of patients whose quality of life was not affected by pain nor by the side effects of medications throughout the follow-up period.
  Adverse effects: the percentage of patients suffering from unresolved side effects from their medications on day 10.

SECONDARY OUTCOMES:
Patient satisfaction, The average number of times patients contacted their physician throughout the follow-up period | 11 days from day 0 (the day of the operation) to day 10 post operation
  Patient satisfaction: the percentage of patients who are satisfied with the medical services on day 10.
  The average number of times patients contacted their physician throughout the follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of pharmacy, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided